CLINICAL TRIAL: NCT01416129
Title: Biomechanical Superiority of Brimless Versus Ischial Ramus Containment (IRC) Sub Atmospheric Transfemoral Interfaces
Brief Title: Southern Bone & Joint Study - Brimless Sockets
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Southern Bone & Joint Specialists, P.A. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 6140101600
Record Dates: First submitted 2011-08-11; First posted 2011-08-12 (Estimated); Results first posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Socket Designs of Transfemoral Amputees.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Comparator: Prosthetic socket standard of care (Active Comparator)
  Interventions: Device: Standard of care socket
- Active Comparator: Prosthetic brimless socket (Active Comparator)
  Interventions: Device: Prosthetic brimless socket

INTERVENTIONS:
Device: Standard of care socket — Amputees' preferred socket.
  Arms: Active Comparator: Prosthetic socket standard of care
Device: Prosthetic brimless socket — Study socket
  Arms: Active Comparator: Prosthetic brimless socket

SUMMARY:
The investigators are comparing a new type of prosthetic socket for above knee amputees to the standard of care. The hypothesis is that the new type of socket will show equivalence to the standard of care using our designated outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transfemoral or knee-disarticulation amputee
* 18 to 85 years of age
* K3 (variable cadence and community) ambulators;
* Be able to independently provide informed consent
* Be willing to comply with study procedures.

Exclusion Criteria:

* History of chronic skin breakdown on the residual limb
* Conditions that would prevent participation and pose increased risk (e.g. unstable cardiovascular conditions that preclude physical activity such as walking)
* Use of any assistive devices/walking aids, beyond a prosthesis, to ambulate
* Unwillingness/inability to follow instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Highsmith, PT,DPT,CP, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care Prosthetic Socket (Ischial Containment): In this crossover study, 5 subjects were randomized to continue using their ischial containment socket socket first. After assessment, subjects crossed over into the other condition.
- Prosthetic Socket (Experimental): Brimless Socket: 5 subjects randomized to the experimental condition then, following assessment, crossed over to accommodate and re-test with the standard of care (ischial containment socket).
Period: Control Condition: Ischial Containment
Arm/Group | Standard of Care Prosthetic Socket (Ischial Containment) | Prosthetic Socket (Experimental): Brimless Socket
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Experimental Condition: Brimless
Arm/Group | Standard of Care Prosthetic Socket (Ischial Containment) | Prosthetic Socket (Experimental): Brimless Socket
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active Comparator: Prosthetic Socket Standard of Care: This socket is the standard of care and is defined by higher trimlines and a medial wall that contains the ischial tuberosity.
- Active Comparator: Prosthetic Brimless Socket: This is the experimental socket condition that includes lower trimlines, below the level of the ischial tuberosity.
- Total: Total of all reporting groups
Arm/Group | Active Comparator: Prosthetic Socket Standard of Care | Active Comparator: Prosthetic Brimless Socket | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (14.7) | 42.9 (14.7) | 42.9 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Gait
Description: Gait will be assessed in terms of biomechanics and spatiotemporal parameters.
Time Frame: Based on preliminary experience with the intervention, accommodation can range from 2 weeks to 3 months. Assessment will be scheduled within 2 weeks following accommodation.
Reporting Status: Not Posted

2. Primary Outcome: Balance and Stability
Description: Balance and stability will be assessed for limits of stability and postural stability.
Time Frame: as for outcome 1
Reporting Status: Not Posted

3. Primary Outcome: Quality of Life
Description: Validated surveys will be used to solicit participants' subjective experience and feedback.
Time Frame: as for outcome 1
Reporting Status: Not Posted

4. Primary Outcome: Socket Pressure
Description: Pressure sensors are placed on the skin and measured.
Time Frame: 10 minutes after fitting with both sockets
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Control Condition: Prosthetic Socket Standard of Care | Active Comparator/Experimental: Prosthetic Brimless Socket
Number analyzed (Participants) | 10 | 10
mm Hg | 841 (600) | 819 (455)

ADVERSE EVENTS:
Arm/Group | Vacuum Assisted Socket | Standard of Care Socket
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No